CLINICAL TRIAL: NCT04534231
Title: Offering Nicotine Patches to All Households in a Municipality With High Smoking Rates: Test of an Idea to Promote Large Increases in Tobacco Cessation
Brief Title: Offering Nicotine Patches to All Households in a Municipality With High Smoking Rates
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Other Study IDs: 122/2019
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Nicotine patch — Nicotine transdermal patches as per product monograph
  Other Names: Nicoderm

SUMMARY:
One municipality with high smoking rates will be selected. A coupon for free-of-charge nicotine patches will be sent to each household. Reductions in the number of people smoking in the chosen municipality from before to after the NRT distribution will be estimated

DETAILED DESCRIPTION:
A coupon offering five weeks of free nicotine patches will be mailed to every household in a small municipality with elevated smoking rates. Up to 800 participants (one per household) will be able to redeem their coupon online or by phone, and receive nicotine patches via postal mail. Participants will be asked to complete a baseline survey containing items relevant to predicting smoking cessation. Participants will be asked to complete a six-month follow-up survey to assess changes in smoking status.

Research Question: Will the concentrated distribution of nicotine patches in a region of high smoking rates lead to large reductions in smoking rates?

ELIGIBILITY:
Inclusion Criteria:

* speak and understand English
* 18 years or older
* smoke 10 or more cigarettes per day for at least 3 months

Exclusion Criteria:

* health contraindications for using nicotine patches without supervision of a doctor (e.g. allergy to tape, pregnant or intending to become pregnant, currently breastfeeding, serious heart or circulation problems not including high blood pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary residents of the target municipality
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
30-day pint prevalence abstinence | 6 months
  No smoking of cigarettes in the past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham JA, Leatherdale ST, Chaiton M, Tyndale RF, Schell C, Godinho A. Concentrated Distribution of Nicotine Patches to a Town With High Smoking Rates-Any Evidence of Large Impacts on Tobacco Cessation? Nicotine Tob Res. 2023 Apr 6;25(5):1060-1061. doi: 10.1093/ntr/ntac244. No abstract available. PMID 36264570
- [Derived] Cunningham JA, Leatherdale ST, Chaiton M, Tyndale RF, Schell C, Godinho A. Offering nicotine patches to all households in a community with high smoking rates: Pilot test of a population-based approach to promote tobacco cessation. Int J Popul Data Sci. 2021 Feb 11;6(1):1400. doi: 10.23889/ijpds.v6i1.1400. PMID 34007899